CLINICAL TRIAL: NCT06831799
Title: ERN-EuroBloodNet European Collaborative Platform to Share COVID-19 Data in Patients With Red Blood Cell Disorders in Real Time
Brief Title: ERN-EuroBloodNet Registry on Patients With Rare Red Blood Cell Defects and COVID-19
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: European Georges Pompidou Hospital (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital Vall d'Hebron (Other); Unidade Local de Saúde de Coimbra, EPE (Other); University Hospital Freiburg (Other); Azienda Ospedaliera di Padova (Other); Hôpital Necker-Enfants Malades (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Erasme University Hospital (Other); Aghia Sophia Children's Hospital of Athens (Other); Cyprus Institute of Neurology and Genetics (Other); University Hospital Heidelberg (Other); Children's Health Ireland (Other Government); San Luigi Gonzaga Hospital (Other); Oxford University Hospitals NHS Trust (Other); UMC Utrecht (Other); General Hospital of Athens Elpis (Other); Amsterdam UMC (Other); Brno University Hospital (Other); Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello (Other); University Hospital, Gentofte, Copenhagen (Other); Institute of Hematology and Blood Transfusion, Czech Republic (Other); Universitaire Ziekenhuizen KU Leuven (Other); Palacky University (Other)
Responsible Party: Sponsor
Other Study IDs: VHI-ERN-2020-00; PR(AG)215/2020 (Other: Ethics Committee Vall d'Hebron Universitary Hospital)
Record Dates: First submitted 2023-02-17; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Hemoglobinopathies; Sickle Cell Disease; Sickle Cell Anemia; Sickle Beta Thalassemia; Sickle-Cell; Hemoglobinopathy; Sickle Cell Hemoglobin C; Sickle Cell Hemoglobin D; Sickle Cell-Hemoglobin E Disease; Beta-Thalassemia; Beta Thalassemia Major; Beta Thalassemia Intermedia; Dominant Beta-Thalassemia; Hereditary Persistence of Fetal Hemoglobin Thalassemia; Delta-Beta Thalassaemia; Haemoglobin C-Beta-Thalassaemia Syndrome; Hemoglobin E-Beta Thalassemia; Alpha-Thalassemia; Hemoglobin H Disease; Hemoglobin Barts Hydrops; Enzyme Disorder; Anemia; Membranes; Disorder; Elliptocytosis, Hereditary; Stomatocytosis; Spherocytosis, Hereditary
Keywords: COVID-19; Hemoglobinopathy; Sickle cell disease; Sickle Cell Anemia; Sickle cell-beta-thalassemia; Sickle cell-hemoglobin; Beta-Thalassemia; Beta Thalassemia Major; Beta Thalassemia Intermedia; Delta-Beta Thalassaemia; Alpha-Thalassemia; Hemoglobin; Rare hemolytic anemia; Hereditary Spherocytosis; Hereditary Elliptocytosis; Hereditary Stomatocytosis
MeSH Terms: conditions — Hemoglobinopathies; Anemia, Sickle Cell; Hemoglobin SC Disease; beta-Thalassemia; Beta Thalassemia, Dominant Inclusion Body Type; Delta-Beta Thalassemia; alpha-Thalassemia; Anemia; Elliptocytosis, Hereditary; Spherocytosis, Hereditary; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (8):
- Pediatric Sickle cell disease patients infected by COVID-19: Sickle cell diagnosed patients (<18 years old) infected by COVID-19
  Interventions: Other: Non applicable, is a patient registry
- Adult Sickle cell disease patients infected by COVID-19: Sickle cell diagnosed patients (≥18 years old) infected by COVID-19
  Interventions: Other: Non applicable, is a patient registry
- Pediatric Thalassemia patients infected by COVID-19: Thalassemia-diagnosed patients (<18 years old) infected by COVID-19
  Interventions: Other: Non applicable, is a patient registry
- Adult Thalassemia patients infected by COVID-19: Thalassemia-diagnosed patients (≥18 years old) infected by COVID-19
  Interventions: Other: Non applicable, is a patient registry
- Pediatric Enzymopathy patients infected by COVID-19: Enzymopathy-diagnosed patients (<18 years old) infected by COVID-19
  Interventions: Other: Non applicable, is a patient registry
- Adult Enzymopathy patients infected by COVID-19: Enzymopathy-diagnosed patients (≥18 years old) infected by COVID-19
  Interventions: Other: Non applicable, is a patient registry
- Pediatric Membranopathy patients infected by COVID-19: Membranopathy-diagnosed patients (<18 years old) infected by COVID-19
  Interventions: Other: Non applicable, is a patient registry
- Adult Membranopathy patients infected by COVID-19: Membranopathy-diagnosed patients (<18 years old) infected by COVID-19
  Interventions: Other: Non applicable, is a patient registry

INTERVENTIONS:
Other: Non applicable, is a patient registry — Non applicable, is a patient registry

SUMMARY:
Patients with red blood cell disorders (RBCDs), such as Sickle cell disease (SCD) and Thalassemia, are chronic, life-threatening conditions that can become multi-organ complications over time, and are likely at an increased risk of COVID-19-related complications. Patients at the highest risk include the elderly (>50 in our population), those with a history of respiratory or cardiac disease and those with other comorbidities. Several patients affected by RBCDs undergo splenectomy as therapeutic option to improve their level of hemoglobin concentration. Splenectomized patients, or in the case of SCD with functional hyposplenism, are more vulnerable to bacterial infections / superinfections after viral infection. Acute pulmonary syndrome (ACS) is the main cause of morbidity in SCD in middle-high income countries, and is often triggered by infectious events. Currently, there is no literature on the subject. Thus, any recommendation available comes from the experience gained with previous Coronaviruses infections. Accordingly, the correct treatment and management of infection by Coronavirus SARS-COV-2 (COVID-19) in patients affected by RBCDs may be challenging given the rapid spread of the pandemic and limited literature so far, especially in some countries. Accordingly, there is an urgent need to pool evidence in a unique repository on patients affected by RBCDs and COVID-19 in order to reach critical numbers to facilitate the medical decision making process across Europe.

The Registry on patients with rare RBCDs and COVID-19 is an initiative conceived in the core of the European Reference Network on Rare Hematological Diseases (ERN-EuroBloodNet, FPA 739541, www.eurobloodnet.eu) aiming at supporting medical practice of COVID-19 in these patients by gathering evidence on pediatric and adult COVID-19 confirmed cases in RBCDs across Europe.

DETAILED DESCRIPTION:
The Registry on patients with rare red blood cell disorders (RBCDs) and COVID-19 is an initiative conceived in the core of the European Reference Network on Rare Hematological Diseases (ERN-EuroBloodNet, FPA 739541, www.eurobloodnet.eu) aiming at supporting medical practice of COVID-19 in these patients by gathering evidence on pediatric and adult COVID-19 confirmed cases in RBCDs across Europe.

Primary objective of the registry is to pool evidence on the clinical management and outcomes of patients affected by red blood cell disorders and COVID-19 for supporting daily medical practice while enabling inter-professional consultation of complex cases. Secondary objective includes the performance of observational studies in the different cohorts of patients, including Sickle Cell Disease, Thalassaemia, Enzymopathies and Membranopathies patients in pediatric and or adult stages.

The network of hospitals that will be created from this registry will hold regular meetings to analyze the data that are being introduced and to discuss possible measures against COVID-19 based on them. The collaboration will continue with the development of observational studies that will give the necessary evidence to make recommendations for COVID-19 management in hematological patients.

METHODOLOGY

Inclusion criteria include both pediatric and adults patients with confirmed COVID-19 and affected by a rare anaemia disorder due to a red blood cell defect. Data set elements include:

* Demographics: country of living, sex, age (only year of birth)
* Data related to Red blood cell disorder: diagnosis, co-morbidities, treatments, splenectomy, blood transfusion requirement.
* Data related to COVID-19: date and method for diagnosis, severity grade, clinical manifestations i.e. pneumonia, symptoms days, acute events, treatments, days of hospitalization, days at intensive care unit, sequela, death.

The registry has been developed by Vall d'Hebron Research Institute using Redcap, a secure web application for building and managing online databases. Individual patients' data will be gathered in a codified way.

ETHICS AND GDPR COMPLIANCE

The processing of personal data is conducted fully respecting the Regulation (EU) 2016/679 (General Data Protection Regulation), including legal basis and special requirements and safeguards to ensure the safety and the confidentiality of the data subjects.

The Research Ethics Committee of the Vall d'Hebron's Hospital has confirmed that this exceptional case justifies the waiver of informed consent.

PROCESSING OF THE DATA

The patient's information included in the database is pseudonymised by single codification. The minimization principle of data protection is followed (i.e. only year of age is collected, no identified data is collected, and only clinical data of the health care is collected). The medical doctors at each center have a coding table in which the code can be linked to the patient's personal information. This table is safely guarded by the medical doctor and never leaves the center. All the information stored in the database is pseudonymised.

ELIGIBILITY:
Inclusion Criteria:

* Patients both pediatric and adults with confirmed COVID-19 and affected by a rare anaemia disorder due to a red blood cell defect

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients both pediatric and adults with confirmed COVID19 and affected by a rare anaemia disorder due to a red blood cell defect according to the following ORPHA codes for rare diseases:
  * 68364 Hemoglobinopathy
  * 275752 Sickle Cell Disease and related diseases
  * 848 Beta-thalassemia
  * 846 Alpha-Thalassaemia
  * 98363 Rare hemolytic anemia
  * 98369 Rare constitutional hemolytic anemia due to an enzyme disorder
  * 98364 Rare constitutional hemolytic anemia due to a red cell membrane anomaly
Sampling Method: Probability Sample
Enrollment: 684 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical Management and Outcomes in Patients with Red Blood Cell Disorders and COVID-19 | Through study completion, an average of 3 years
  • COVID-19 clinical manifestations and required treatment in each cohort (Sickle Cell Disease, Thalassemia, Enzymopathies, and Membranopathies)..

SECONDARY OUTCOMES:
Secondary Analysis in Different Cohorts of Patients with Red Blood Cell Disorders and COVID-19: | Through study completion, an average of 3 years
  * Descriptive analysis of demographic and baseline disease characteristics in each cohort (Sickle Cell Disease, Thalassemia, Enzymopathies, and Membranopathies).
  * COVID-19 clínical manifestations in each cohort.
  * Identification of preventive measures and risk factors related to severe COVID-19 in each cohort

CONTACTS AND LOCATIONS:
Overall Officials: María del Mar Mañú Pereira, PhD, Principal Investigator — Vall d'Hebron Institut de Recerca, Barcelona (Spain) and ERN-EuroBloodNet; Pablo Velasco Puyó, MD, Principal Investigator — Vall d'Hebron University Hospital, Barcelona (Spain)
Locations (1):
- Vall d'Hebron Institut de Recerca, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Registry platform — https://eurobloodnet.eu/covid/access-to-the-platform/
- See also: ERN-EuroBloodNet Collaborative Platform on Red Blood Cell and COVID-19 patients section — https://eurobloodnet.eu/covid/about-the-platform/
- See also: ERN-EuroBloodNet website — https://eurobloodnet.eu/
- See also: European Commission website section on European Reference Networks — https://health.ec.europa.eu/european-reference-networks/overview_en
- See also: Directive 95/46/EC of the European Parliament and of the Council of 24 October 1995 on the protection of individuals with regard to the processing of personal data and on the free movement of such data — https://eur-lex.europa.eu/legal-content/en/TXT/?uri=CELEX%3A31995L0046